# The GlaxoSmithKline group of companies

205767

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for a randomized, repeat dose, open label, parallel group, multi-center study to evaluate the effect of daprodustat compared to darbepoetin alfa on forearm blood flow in participants with anemia of chronic kidney disease that are not dialysis dependent |
| <b>Compound Number</b> | : | GSK1278863 |
| <b>Effective Date</b> | : | Refer to Document Date |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol GlaxoSmithKline Document Number 2016N291495\_02.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Author | Date |
|---|---|
| Lead | |
| Manager-Statistics (Speciality), Development Biostatistics India Stats | Refer to Document<br>Date |
| <b>Co-Authors</b> | |
| Statistician (Speciality), Development Biostatistics | 02-NOV-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

205767

# **RAP Team Review Confirmations** (Method: E-mail)

| Reviewer | Date |
|---|---|
| PPD (C : 1'(-) D 1 (D: -(-)' (C - 1 1') | 31-OCT-2020 |
| Lead Programmer (Speciality), Development Biostatistics India<br>Prog | 31-001-2020 |
| PPD | |
| Director Clinical Development (Clinical Science Nephrology)<br>Clinical Sciences Respiratory and Specialty | 02-NOV-2020 |
| PPD | |
| Statistics Director (Speciality), Development Biostatistics | 31-OCT-2020 |
| PPD | |
| Global Clinical Development Manager (R&D GCSD),<br>Development Global Clinical Operations | 31-OCT-2020 |
| PPD | |
| Principal Clinical Data Manager (RD PCPS GCDO DM FPD),<br>Development Global Clinical Operations | 02-NOV-2020 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date | Approval<br>Method |
|---|---|---|
| Manager- Statistics (Speciality), Development<br>Biostatistics India Stats | Refer to Document Date | E-signature,<br>eTMF |
| Senior Manager - Programming (Speciality), Development Biostatistics India Prog | Refer to Document Date | E-signature,<br>eTMF |

# **TABLE OF CONTENTS**

# **PAGE**

| 1. | INTRO | DDUCTION | 5 |
|---|---|---|---|
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s). Study Design Statistical Hypotheses. | 5<br>6 |
| 3. | PLANI<br>3.1.<br>3.2. | NED ANALYSES Interim Analyses Final Analyses | 9 |
| 4. | ANALY<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS Study Treatment & Sub-group Display Descriptors Baseline Definitions Multicentre Studies. Other Considerations for Data Analyses and Data Handling Conventions | 10<br>11 |
| 6. | STUD'<br>6.1.<br>6.2. | Overview of Planned Study Population Analyses Display Details 6.2.1. Study Disposition 6.2.2. Protocol Deviations 6.2.3. Demographic and Baseline Characteristics 6.2.4. Medical Conditions, Prior and Concomitant Medications 6.2.5. Exposure | 12<br>12<br>12<br>13<br>13 |
| 7. | 7.1.<br>7.2. | TY ANALYSES Adverse Events Analyses Clinical Laboratory Analyses Other Safety Analyses | 14<br>14 |
| 8. | PHAR 8.1. | Primary Pharmacodynamic Analyses 8.1.1. Endpoint / Variables 8.1.2. Summary Measure 8.1.3. Population of Interest 8.1.4. Strategy for Intercurrent (Post-Randomization) Events 8.1.5. Statistical Analyses / Methods Secondary Pharmacodynamic Analyses | 15<br>16<br>16<br>16 |
| | 0.2. | 8.2.1. Endpoint / Variables | 16 |

205767

| | | 8.2.4.<br>8.2.5. | Strategy for Intercurrent (Post-Randomization) Events | |
|---|---|---|---|---|
| 9. | REFER | RENCES. | | 18 |
| 10 | 4 DDEN | IDIOEC | | 40 |
| 10. | | | (1. Protocol Deviation Management and Definitions for Dev | 19 |
| | 10.1. | | 1: Protocol Deviation Management and Definitions for Per Population | 10 |
| | | | Exclusions from Per Protocol Population | |
| | 10.2. | Δnnendiy | 2: Schedule of Activities | 20 |
| | 10.2. | | Protocol Defined Schedule of Activities | |
| | 10.3. | | 3: Assessment Windows | |
| | 10.0. | | Definitions of Assessment Windows for Analyses | |
| | 10.4. | | 4: Study Phases and Treatment Emergent Adverse | 20 |
| | . • | | | 24 |
| | | 10.4.1. | Study Phases | |
| | | | 10.4.1.1. Study Phases for Concomitant Medication | |
| | | 10.4.2. | Treatment Emergent Flag for Adverse Events | |
| | 10.5. | Appendix | c 5: Data Display Standards & Handling Conventions | |
| | | 10.5.1. | Reporting Process | |
| | | 10.5.2. | Reporting Standards | 25 |
| | 10.6. | Appendix | c 6: Derived and Transformed Data | 27 |
| | | 10.6.1. | General | 27 |
| | | 10.6.2. | Study Population | 27 |
| | | 10.6.3. | Safety | |
| | | 10.6.4. | Pharmacodynamic | |
| | 10.7. | Appendix | 7: Reporting Standards for Missing Data | |
| | | 10.7.1. | Premature Withdrawals | |
| | | 10.7.2. | Handling of Missing Data | |
| | | | 10.7.2.1. Handling of Missing and Partial Dates | |
| | 10.8. | | (8: Values of Potential Clinical Importance | |
| | | 10.8.1. | Laboratory Values | |
| | | 10.8.2. | Vital Signs | |
| | | 10.8.3. | FBF | |
| | 40.0 | 10.8.4. | PWV | |
| | 10.9. | | ( 9: Abbreviations & Trademarks | |
| | 40.40 | | Trademarks | |
| | 10.10. | | ( 10: List of Data Displays | |
| | | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| | | 10.10.5. | Safety Tables Pharmacodynamic Tables | 30 |
| | | | ICH Listings | |
| | | | Non-ICH Listings | |
| | 10 11 | | (11: Example Mock Shells for Data Displays | |
| | | pponal/ | | ***** |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol GlaxoSmithKline Document Number 2016N291495 02.

| Revision Chronology: | | |
|---|---|---|
| Protocol number: | Date: | Version: |
| 2016N291495_00 | 17/Nov/2017 | Original Protocol |
| 2016N291495_01 | 28/Jan/2018 | Protocol Amendment 1 |
| This protocol amendment was written as the study team was required per regulatory agencies to change the protocol to include serum pregnancy testing at screening. During the amendment process, minor updates were made for study optimization. | | |
| 2016N291495_02 | 07/Aug/2019 | Protocol Amendment 2 |
| This protocol amendment was written becase a challenge agent suddenly became commercially unavailable with no immediate ability to reobtain this. The study has been modified to allow flexibility for the forearm blood flow testing to be performed with this agent if it becomes available again, and to be performed without it if not. | | |
| During this time the safe | ety language was updated a | s well. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| 10.1.2 Sample Size Re-<br>estimation | Sample size re-estimation<br>will not be performed | The study was terminated |
| 10.3.3 Other Analyses<br>(Pharmacodynamic) | No statistical analyses will<br>be performed; only<br>summary statistics will be<br>reported. We will not<br>perform exploratory<br>analyses and sensitivity<br>analysis. | Since the study was terminated and we have only 4 completed subjects to report. Therefore, statistical analysis will not be performed. |

205767

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| 10.3.4 Interim Analyses | Interim analyses will not be<br>performed | The study was terminated |
| Enrolled population is not defined in the protocol | <ul> <li>Enrolled population added<br/>in the RAP with the below<br/>definition.</li> <li>"All Randomized<br/>Participants"</li> </ul> | This population is required for data disclosure displays |
| 10.2. Pharmacodynamic Per-Protocol (PDPP) Population: "All randomized participants who provide pharmacodynamic (PD) data at Day 1 and Day 42 that meets the QC criteria (See Section 9.6.1.3 of Protocol) and completes the protocol without important deviations will be included in the PDPP population. This population will be used in the evaluation of all endpoints with the exception of safety endpoints." | PDPP definition updated with adding RAP section number of exclusions of per proptocol population. "All randomized participants who provide pharmacodynamic (PD) data at Day 1 and Day 42 that meets the QC criteria (See Section 9.6.1.3 of Protocol) and completes the protocol without important deviations (exclusions are populated under Section 10.1.1 of RAP) will be included in the PDPP population. This population will be used in the evaluation of all endpoints with the exception of safety endpoints." | To exclude all participants based on the Protocol Deviation Management Plan (PDMP) definitions, as not all important deviations are criticial for analysis population exclusion. In efforts to maximize the number of participants in the analysis, only the important deviations (exclusions are populated under Section 10.1.1 of RAP) will be considered exclusionary for the analysis. |
| Non-Contact, Optical Forearm<br>Plethysmography (NC-OFP)<br>Sub-Study | Sub-study will not be performed | The study was terminated,<br>and no subjects recruited<br>for sub-study |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objective | Primary Endpoint |
| To compare the effect of daprodustat to darbepoetin alfa on endothelial function | Change in FBF ratio from Day 1 to Day 42 in response to acetylcholine |
| Principle Secondary | Principle Secondary Endpoint |
| To further compare the effect of daprodustat to darbepoetin alfa on endothelial function | Change in the absolute FBF from Day 1 to Day 42 in response to acetylcholine |
| Secondary Objectives | Secondary Endpoints |
| To compare the effect of daprodustat to darbepoetin alfa on endothelium-independent vasodilation | Change in FBF ratio from Day 1 to 42 in response to sodium nitroprusside (SNP) |

205767

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Change in the absolute FBF from Day 1 to Day 42 in response to SNP</li> </ul> |
| To compare the effect of daprodustat to darbepoetin alfa on basal endothelial NO synthesis | <ul> <li>Change in FBF ratio from Day 1 to Day 42 in response to L-N<sup>G</sup>-monomethyl arginine citrate (L-NMMA)</li> <li>Change in the absolute FBF from Day 1 to Day 42 in response to L-NMMA</li> </ul> |
| To compare the effect of daprodustat on the FBF response to acetylcholine, SNP and L-NMMA between Day 42 and Day 1 | <ul> <li>Change in FBF ratio in response to each individual challenge agent at Day 42 vs Day 1 in participants treated with daprodustat</li> <li>Change in the absolute FBF in response to each individual challenge agent at Day 42 vs Day 1 in participants treated with daprodustat</li> </ul> |
| To compare the effect of darbepoetin alfa on the FBF response to acetylcholine, SNP and L-NMMA between Day 42 and Day 1 | <ul> <li>Change in FBF ratio in response to each individual challenge agent at Day 42 vs Day 1 in participants treated with darbepoetin alfa</li> <li>Change in the absolute FBF in response to each individual challenge agent at Day 42 vs Day 1 in participants treated with darbepoetin alfa</li> </ul> |
| To compare the effect of daprodustat to darbepoetin alfa on vascular compliance | Change in Augmentation Index (an indicator of arterial stiffness) as estimated by radial arterial pulse contours from Day 1 to 42 Change in pulse wave velocity (PWV) from Day 1 to Day 42 |
| Safety | Safety Endpoints |
| Assess safety and tolerability | <ul> <li>Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) including AEs of special interest</li> <li>Reasons for discontinuation of randomized study treatment</li> <li>Absolute values and changes from baseline in clinical laboratory parameters, ECG parameters, blood pressure (BP) and heart rate (HR)</li> </ul> |
| Exploratory Objective | Exploratory Endpoint |
| To explore the relationship between diabetes status and endothelial function | <ul> <li>FBF response to each individual challenge agent in relation to diabetes status</li> </ul> |

# 2.3. Study Design



# 2.4. Statistical Hypotheses

The primary endpoint is to compare the effect of daprodustat to darbepoetin alfa on change in FBF ratio from Day 1 to Day 42 in response to acetylcholine. The estimand of interest is the effect of 6 weeks of randomized treatment on the primary endpoint.

**Null:** The difference between daprodustat and darbepoetin alfa on the acetylcholine-induced change (from Day 1) in FBF ratio at Day 42 is 0.

**Alternative:** The difference between daprodustat and darbepoetin alfa on the acetylcholine-induced change (from Day 1) in FBF ratio at Day 42 is not 0.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

The study was terminated, hence no interim analysis will be performed.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed an ICF to participate in<br>the clinical trial. This population will be used for<br>summarizing screening failure rates and reasons for<br>screening failure. | Screen Failures |
| Safety | <ul> <li>All randomized participants who receive at least one dose of study treatment will be included in the safety population.</li> <li>This population will be used in the evaluation of all safety analyses</li> <li>Participants will be analyzed according to the treatment received.<sup>1</sup></li> </ul> | <ul><li>Study population</li><li>Safety and tolerability</li></ul> |
| Pharmacodynamic<br>Per-Protocol<br>(PDPP)<br>Population | All randomized participants who provide pharmacodynamic (PD) data at Day 1 and Day 42 that meets the QC criteria (See Section 9.6.1.3 of Protocol) and completes the protocol without important deviations (exclusion are populated under | Primary,<br>secondary<br>endpoints |

205767

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | Section 10.1.1 of RAP) will be included in the PDPP | |
| | population. | |
| | This population will be used in the evaluation of all | |
| | endpoints with the exception of safety endpoints. | |
| | <ul> <li>Participants will be analyzed according to the</li> </ul> | |
| | treatment received.1 | |
| Enrolled | All randomized participants | <ul> <li>Study population</li> </ul> |

<sup>[1]:</sup> Only participants receiving incorrect randomized treatment for the duration of their study participation will be analysed according to the treatment received. Otherwise, participants will be analyzed according to the treatment to which they were randomized.

Refer to Appendix 10: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [28Aug2018 V2.0].

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG System Data Displays for Reporting | | | |
| Code | Description | Description | Order in TLF |
| А | Darbepoetin alfa | rhEPO | 2 |
| В | Daprodustat | Dapro | 1 |

## 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Primary Endpoint | | | | |
| FBF ratio | | | X | Day 1/Repeat Day 11 |
| Secondary Endpoints | | | | |
| FBF ratio | | | X | Day 1/Repeat Day 11 |
| Absolute FBF | | | X | Day 1/Repeat Day 11 |
| Augmentation index | | | X | Day 1/Repeat Day 11 |
| PWV | | | X | Day 1/Repeat Day 11 |
| Clinical laboratory<br>parameters, ECG<br>parameters, blood<br>pressure (BP) and<br>heart rate (HR) | X | | X | Screening/Day 1 |

<sup>&</sup>lt;sup>1</sup>Repeat Day 1 values are only used if a repeat visit was deemed necessary

Unless otherwise stated, if baseline data is missing, no derivation will be performed, and baseline will be set to missing. If a Repeat Day 1 visit is required, then this value will be used as the baseline measurement instead.

## 5.3. Multicentre Studies

Participants will be recruited from 3 centers and will be randomised stratifying by centre. Enrolment will be presented by investigative site.

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Screened/Enrolled/Safety population, unless otherwise specified. The study population analyses will include a total column, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards.

Details of the planned displays are presented in Appendix 10 List of Data Displays.

# 6.2. Display Details

# 6.2.1. Study Disposition

## Participant Status and Reason for Study Withdrawal

The number and percentage of subjects who completed the study as well as participants who withdrew from the study will be summarized by participant status and reason for withdrawal. Also, a summary of number of subjects by country and site id by treatment group and overall total.

A listing of reasons for study withdrawal will be provided for all participants who were withdrawn from the study.

## Screening Status and Reasons for Screen Failure

The number and percentage of participants who passed screening (i.e. enrolled) and who failed screening and therefore were not entered into the study will be summarized along with the reasons for failure will be summarized for those participants who failed screening. If a subject has been screened multiple times, the subject's latest screening information will be displayed. (Note that the reasons for rescreened participants who initially failed but subsequently enrolled are not included in the display.)

A listing of the screen failure record for all participants who failed screening and were not enrolled in the study will be produced. This listing will include site ID, unique subject ID, date of screen failure, reason term(s) for screen failure (including the specify text, if any).

## 6.2.2. Protocol Deviations

A listing of important protocol deviations will be provided. The listing will include treatment, site ID, unique subject ID, date of deviation, study day of deviation, protocol deviation category, protocol deviation coded term, and protocol deviation description.

205767

A listing of participants with inclusion/exclusion criteria deviations will be provided. The listing will include treatment, site ID, unique subject ID, inclusion/exclusion type, and criteria description.

## 6.2.3. Demographic and Baseline Characteristics

## <u>Demographic Characteristics</u>

Demographic data will be summarized by treatment group and overall.

A listing of demographic and baseline characteristics will also be produced. This listing will include treatment, site ID, unique subject ID, year of birth, age, sex, ethnicity, height, weight, and other demographic and baseline characteristics.

## <u>Age Ranges</u>

A summary of age ranges will be produced for each treatment group and overall total.

## Race and Racial Combinations

A summary of race and racial combinations will be produced for each treatment group and overall total.

# 6.2.4. Medical Conditions, Prior and Concomitant Medications

## Medical Conditions

A listing of medical conditions will be produced, which will capture both pre-specified medical conditions and other medical conditions collected on the eCRF.

## Concomitant Medications

A listing of all medications taken by participants, including any of which are pre, on and post-treatment, will be produced. The relationship between ATC level 1, 2, 3, and ingredients and verbatim text for all medications in the study will be listed.

## 6.2.5. Exposure

A listing of exposure data will be provided. This listing will include treatment, site ID, unique subject ID, dose start date, duration of time on dose, dose and dose units.

## 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

| Objectives | Endpoints |
|---|---|
| Safety | |
| Assess safety and tolerability | <ul> <li>Incidence and severity of adverse events<br/>(AEs) and serious adverse events (SAEs)<br/>including AEs of special interest</li> </ul> |
| | <ul> <li>Reasons for discontinuation of randomized<br/>study treatment</li> </ul> |
| | <ul> <li>Absolute values and changes from baseline<br/>in clinical laboratory parameters, ECG<br/>parameters, blood pressure (BP) and heart<br/>rate (HR)</li> </ul> |

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

Adverse Events

A listing of AE records for all participants who reported AEs will be produced.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays and include the following tests:

205767

| Laboratory<br>Assessments | Parameters | | |
|---|---|---|---|
| | Platelet count | RBC indices: | WBC count with<br>Differential |
| | RBC count | MCV | Neutrophils |
| Hematology | Reticulocyte count | MCH | Lymphocytes |
| | Hgb | MCHC | Monocytes |
| | Hematocrit | RDW | Eosinophils |
| | WBC count (Absolute) | | Basophils |
| | Sodium (serum) | AST <sup>1</sup> | Carbon Dioxide (total) |
| | Potassium (serum) | ALT <sup>1</sup> | Albumin |
| Clinical Chemistry <sup>1</sup> | Creatinine (serum) | Chloride (serum) | Urea (serum) |
| | Glucose | Bilirubin (total and | Alkaline Phosphatase |
| | | direct/indirect) | |
| | Serum ferritin | TSAT | hs-CRP |
| | Total cholesterol | LDL-C (direct) | HDL-C |
| | Triglycerides | Serum/Urine hCG | FSH <sup>3</sup> |
| | | pregnancy test <sup>2</sup> | |
| Other laboratory tests | HbA1c | Folate | Vitamin B <sub>12</sub> |
| | Serology (hepatitis B | | |
| | surface antigen | | |
| | [HBsAg], and hepatitis | | |
| | C virus antibody) | | |

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

# 8. PHARMACODYNAMIC ANALYSES

# 8.1. Primary Pharmacodynamic Analyses

# 8.1.1. Endpoint / Variables

The endpoint of interest is FBF ratio.

FBF ratio is calculated as the FBF of the subject's treatment arm divided by the subject's non-treatment arm. The treatment arm is given either saline or the challenge agent. The non-treatment arm is given nothing.

The FBF measurement is calculated from the average of 5 values as recorded on the LabChart file. The 5 values of FBF are recorded manually from a blinded central reader reviewing the subject's FBF LabChart file.

## 8.1.2. Summary Measure

The summary measure of interest is the change in FBF ratio from Day 1 to Day 42 in response to acetylcholine.

If FBF procedure is repeated for Day 1 and/or Day 42, this data will take the place of the original Day 1 and Day 42 data respectively. A quality control (QC) check will be performed on the FBF data before the final analyses. The QC check will be to assess negative and extreme values for FBF (FBF).

Descriptive statistics (n, arithmetic mean, standard deviation (SD), minimum, median, maximum) will be calculated by treatment group for change in FBF ratio endpoints.

## 8.1.3. Population of Interest

The primary pharmacodynamics analyses will be based on the PDPP population, unless otherwise specified.

# 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Due to the design of the PDPP population, only subjects who have FBF measurements for both Day 1 and Day 42 are included, and it is not possible to have missing FBF data. Therefore, no FBF data will be imputed.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics and listed.

# 8.2. Secondary Pharmacodynamic Analyses

## 8.2.1. Endpoint / Variables

- Principle secondary endpoint: change in the absolute FBF
- Secondary endpoints:
  - o FBF ratio, absolute FBF of Sodium nitroprusside and L-NMMA
  - Augmentation index
  - o PWV

Absolute FBF is defined as only including the FBF value from the subject's treatment arm which is infused with either saline or challenge agents.

## 8.2.2. Summary Measure

Principle secondary endpoint: Change in the absolute FBF from Day 1 to Day 42 in response to acetylcholine

Secondary endpoints: Change in FBF ratio from Day 1 to Day 42 in response to sodium nitroprusside and L-NMMA.

Change in absolute FBF from Day 1 to Day 42 in response to sodium nitroprusside and L-NMMA.

Change in Augmentation Index (AIX, an indicator of arterial stiffness) as estimated by radial arterial pulse contours from Day 1 to Day 42.

Change in pulse wave velocity (PWV) from Day 1 to Day 42.

For the PWV dataset, there are two recorded values for each variable per day, with the option to collect a third value if the first two values varied (Refer: SRM) too much from each other. The average of the two closest absolute values will be used for analysis purposes.

If for any of these measures mentioned above, the respective procedures are repeated for Day 1 and/or Day 42, the data from the repeat visit will take place of the original Day 1 and Day 42 data respectively. Like the FBF data, a QC check will be performed for the PWV data before the final analyses. The QC check will be to assess negative and extreme values for PWV (PWV).

Descriptive statistics (n, mean, standard deviation (SD), minimum, median, maximum) will be calculated by treatment group.

## 8.2.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the PDPP population, unless otherwise specified.

## 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

Augmentation index and PWV data is expected to have minimal missing data, therefore these data points will not be imputed if missing.

## 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10 List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics and listed.

205767

# 9. REFERENCES

- GlaxoSmithKline Document Number 2016N291495\_02. A randomized, repeat dose, open label, parallel group, multi-center study to evaluate the effect of daprodustat compared to darbepoetin alfa on forearm blood flow in participants with anemia of chronic kidney disease that are not dialysis dependent; 07-Aug-2019.
- GUI 137354: Information for Authors Reporting and Analysis Plan, Global; GSK.
- Iverson C, Christiansen S, Flanagin A, et al. AMA Manual of Style: A Guide for Authors and Editors. 10th ed. New York, NY: Oxford University Press; 2007.
- Medicines and Healthcare Products Regulatory Agency. Recombinant human erythropoietins: New advice for prescribing. Drug Safety Update. 2007; 1:2.
- SOP\_54838: Development, Review & Approval of Reporting & Analysis Plan, Global; GSK.

205767

# 10. APPENDICES

# **10.1.** Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 10.1.1. Exclusions from Per Protocol Population

There is no important protocol deviation identified in the study, hence no exclusions for per protocol population.

205767

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Activities

| | Screening <sup>1</sup> | | | Treatme | nt Period² | | | Follow-up <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|
| Procedure | Up to 30 Days | Day 1 | Repeat<br>Day 1 <sup>17</sup> | Day 14 | Day 28 | Day 42 | Repeat<br>Day 42 <sup>17</sup> | |
| Informed consent | X | | | | | | | |
| Eligibility Criteria | X | X <sup>4</sup> | | | | | | |
| Physical examinations, Medical History, Demographics | Х | <b>X</b> <sup>5</sup> | | | | | | |
| HemoCue Hgb | X | X6 | Х | Χ | Х | Х | Х | |
| eGFR | Х | | | | | | | |
| Vital signs | X | X6 | Х | Χ | Х | Х | Х | Χ |
| Clinical chemistry <sup>7</sup> | Х | | | | | Х | | Χ |
| Hematology <sup>7</sup> | Х | Х | | Χ | Х | Х | | Х |
| Serum pregnancy test (FRP only) | Х | | | | | | | |
| Urine pregnancy test (FRP only)8 | | Х | Х | Χ | Х | Х | Х | Х |
| Folate & Vitamin B <sub>12</sub> | Х | | | | | | | |
| 12 Lead ECG | X | X6 | | | | Х | | Χ |
| Ferritin & TSAT | Х | | | | | | | |
| hs-CRP | Х | Х | | | | Х | | |
| Females only: FSH <sup>9</sup> | Х | | | | | | | |
| 5Brachial artery palpation | X | | | | | | | |
| Randomization | | Х | | | | | | |
| Daprodustat administration <sup>10</sup> | | <===== | ======= | ======== | | ======== | ====> | |
| Darbepoetin alfa administration <sup>10</sup> | | | (10 | X | Х | See<br>footnote<br>18 | | |

205767

| | Screening <sup>1</sup> | Treatment Period <sup>2</sup> | | | | | Follow-up <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|
| Procedure | Up to 30 Days | Day 1 | Repeat<br>Day 1 <sup>17</sup> | Day 14 | Day 28 | Day 42 | Repeat<br>Day 42 <sup>17</sup> | |
| Study treatment adjustment <sup>11</sup> | | | | | Χ | | - | |
| Liver chemistry monitoring | | | | Χ | Χ | | | |
| International Normalized Ratio (INR)12 | Х | Χ | Χ | | | Х | Х | |
| Hepatitis B and C screening <sup>13</sup> | Х | | | | | | | |
| HbA1c, lipids <sup>7</sup> | | Χ | | | | | | |
| Forearm Blood Flow (FBF)14 | | Χ | Χ | | | Х | Х | |
| Pulse Wave Velocity (PWV) <sup>14</sup> | | Χ | Χ | | | Х | Х | |
| AE and SAE Assessment | X <sup>15</sup> | Χ | Χ | Х | Χ | Х | Х | Х |
| Blood draw for storage biomarkers <sup>16</sup> | | Χ | | | | Х | | |
| Review concomitant medications | Х | Χ | Х | Х | Χ | Х | Х | Х |

<sup>&</sup>lt;sup>1</sup> All participants will undergo screening assessments within 30 days of enrolment.

<sup>&</sup>lt;sup>2</sup> Allowable time window  $\pm$  2 days except for the forearm blood flow (FBF) & pulse wave velocity (PWV) as noted.

<sup>&</sup>lt;sup>3</sup> Allowable time window ± 3 days. Follow up will occur 7-14 days ± 3 following completion of the last FBF procedure. See Section 8.2 for guidance regarding EW participants.

<sup>&</sup>lt;sup>4</sup> Eligibility criteria to be assessed prior to performance of the FBF procedure include HemoCue hemoglobin (Hgb), vital signs & 12-lead electrocardiogram (ECG).

<sup>&</sup>lt;sup>5</sup>Only a brief physical exam on Day 1.

<sup>&</sup>lt;sup>6</sup> As detailed in Exclusion Criteria (Section 6.2).

<sup>&</sup>lt;sup>7</sup> Clinical chemistry, hematology and other laboratory tests as listed in Appendix 2.

<sup>&</sup>lt;sup>8</sup>Local urine pregnancy testing will be standard for protocol unless serum testing is required by local regulations or Institutional Review Board (IRB)/ Independent Ethics Committee (IEC).

<sup>&</sup>lt;sup>9</sup> As detailed in Inclusion Criteria (Section 6.1).

<sup>&</sup>lt;sup>10</sup> The initial dose of study treatment will be **after** the Day 1/Repeat Day 1 FBF & PWV procedures. Participants will receive **EITHER** daprodustat **OR** darbepoetin alfa. The final dose of darbepoetin alfa will be Day 41 (i.e., the day prior to the FBF & PWV procedures), while the final dose of darbepoetin alfa will be Day 28. If repeat procedures are needed the dosing will be extended (See Section 9.6.1.4).

205767

<sup>&</sup>lt;sup>11</sup> See Section 7.2 for details on study treatment adjustment

<sup>&</sup>lt;sup>12</sup> Applies only to participants on anti-coagulant therapy; further details concerning measurement of the international normalised ratio (INR) and subsequent actions can be found in the study reference manual (SRM).

<sup>&</sup>lt;sup>13</sup> If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required

<sup>&</sup>lt;sup>14</sup>The FBF & PWV assessments are to be performed following confirmation of INR < 3.0 for participants on anticoagulant therapy. The Day 42 FBF & PWV assessments can be delayed up to 1 week (i.e., Day 49)., while randomization (Day 1) should be delayed until the participant's INR < 3.0 (Section 9.6.1.1).

<sup>&</sup>lt;sup>15</sup>Only serious adverse events (SAEs) assessed as related to study participation are collected at this visit. See Appendix 4 for additional details.

<sup>&</sup>lt;sup>16</sup> As described in Section 9.8

<sup>&</sup>lt;sup>17</sup>Indicates the procedures to be performed on the repeat visits only if the visit is deemed necessary. See Section 9.6.1.4.

<sup>&</sup>lt;sup>18</sup>Darbepoetin is only to be given on Day 42 if a Repeat Day 42 is needed.

205767

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Assessment Windows for Analyses

Data for continuous variables will be summarized according to the scheduled visit time period for which they were recorded in the eCRF. Unscheduled assessments will not be slotted to a particular time point but will remain as unscheduled if they are either summarized or listed unless otherwise specified.

# **10.4.** Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start and stop dates.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 1 day |
| Post-Treatment | Date > Study Treatment Stop Date + 1 day |

• If the treatment stop date is missing and the treatment start date is non-missing, then the assessment will be considered On-Treatment.

## 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

## NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date + 1 day</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 1 day.</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Reporting Process

| Software | |
|---|---|
| The SAS Version 9.4 or above will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound : arenv/arprod/ GSK1278863/mid205767/final_01 | |

## **Analysis Datasets**

- Analysis datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) standards: Study Data Tabulation Model (SDTM) implementation guide (IG) Version 3.1.3 with some updates from Version 3.2, Analysis data model (ADaM) IG Version 1.1, and GSK ADaM specification template.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from system independent (SI) to SDTM.

#### **Generation of RTF Files**

• Rich text format (RTF) files will be generated for Tables

# 10.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- In all displays (TFLs) the term "Subjects" will be used to refer to the "Participants".

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

## Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:

205767

| Statistical Pri | <ul> <li>Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL<br/>Statistical Principle 5.05.1).</li> </ul> |
|---|---|
| <ul> <li>Unscheduled</li> </ul> | or unplanned readings will be presented within the subject's listings. |
| Unscheduled Visits | |
| <ul> <li>Unscheduled visit</li> </ul> | s will not be included in summary tables and/or figures. |
| All unscheduled v | isits will be included in listings. |
| Descriptive Summary | y Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Sta | tistical Principals 7.01 to 7.13. |
| Note | |
| All displays (TFL) will use the term 'Subjects' (i.e. reflect GSK Display Standards and CDISC SDTM/ADaM standards) | |

205767

# 10.6. Appendix 6: Derived and Transformed Data

## 10.6.1. **General**

## Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values for time points other than the baseline within a time window (as per Section 10.3.1), the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.

## Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## **Screening and Washout visits**

• Rescreened subject's data will only be counted once, the latest visit will only be summarized.

# 10.6.2. Study Population

## **Demographics**

## Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)]2

## **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula: The study
  duration will be assigned based on exposure date and by default will assign as 1 day for each date (if
  there is any repetation in the date we will consider only one record). Since there is no exposure end
  date collected for the study, we will be assigning by default value as 1 day. However, we are
  checking duplication in the bakend.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula: Sum of each record in incremental order on all previous records and current record value get added as cumulative.
- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

# 10.6.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</p>

## **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '≤x' or '≥x' is present, then the corresponding numeric value will be set equal to x.
- If there is more than one laboratory value on the same date for the same laboratory test, then the laboratory values associated with scheduled visits will be used.
- The following will be used to convert laboratory values from SI units to conventional units if the specific lab value is not already in this format. [Iverson, 2007]:
  - Hemoglobin and MCHC: Divide the g/L value by 10 to get the g/dL value.
  - TSAT: If unit is not percentage then multiply with 100 to get the % value.
- Lab values that are converted will be reported in place of original value
- Heart rate and pulse rate can be used interchangeably
- Total calcium and calcium can be used interchangeably
- Total protein and protein can be used interchangeably
- Total bilirubin and bilirubin can be used interchangeably
- TSAT and transferrin saturation can be used interchangeably
- Folate and Vitamin B9 can be used interchangeably
- Baseline HGB will be based either on the pre-dose value on Day 1 or screening value. Any
  unscheduled HGB values taken after the pre-dose value on Day 1 will not be used.
- Scheduled central laboratory HGB values and HemoCue HGB value will be used for report.
   Conversion values (g/L value g/dL) also will be reported.

# **PCI Criteria Categories**

- PCI criteria categories are: To Low, To w/in Range or No Change, To High
- Subjects with a missing baseline value are to be assumed to have a normal/within range baseline value.

# 10.6.4. Pharmacodynamic

## Primary/Principle Secondary/Secondary/Exploratory Endpoints

## FBF Ratio/Absolute FBF

- If either a Day 1 Repeat or Day 42 Repeat measurement is available for forearm blood flow, the repeat value will be used instead.
- Forearm blood flow for a given challenge agent dose (infused arm), or for values from the noninfused arm, will be the mean of 5 continuous time point values.
- Forearm blood flow ratio is defined as the ratio of a subject's treatment (infused) arm value divided by the non-treatment (non-infused) arm value
  - First, the mean of both the infused and non-infused arm will be taken separately for the given five measurements before going into the ratio calculation. An example of this is shown in the table below:

205767

| Primary/Principle Secondary/Secondary/Exploratory Endpoints | | | | |
|---|---|---|---|---|
| | | Infused | Non-Infused | |
| | Measurement 1 | 1.2 | 1.01 | |
| | Measurement 2 | 1.1 | 1 | |
| | Measurement 3 | 1.4 | 1.2 | |
| | Measurement 4 | 1.5 | 1.1 | |
| | Measurement 5 | 1.6 | 1.3 | FBF Ratio |
| | Average | 1.36 | 1.122 | 1.212121212 |
| Absolute for | Absolute forearm blood flow is defined as the infused arm value. | | | |

# **Secondary Endpoint**

# **PWV Dataset**

For the PWV dataset, there are two recorded values for each variable per day, with the option to collect a third value if the first two values varied (Refer: SRM) too much from each other. The average of the two closest absolute values will be used for analysis purposes.

# 10.7. Appendix 7: Reporting Standards for Missing Data

# 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as a participant who has completed all phases of the study including the last visit or the last scheduled procedure |
| | Withdrawn subjects were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields<br/>on the collection instrument:</li> </ul> |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing and Partial Dates

| Reporting Detail |
|---|
| Partial dates will be displayed as captured in subject listing displays. |
| <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> <li>Missing Start Month: 'January' will be used unless this makes the start date before the month of start of study treatment; in this case the month of study treatment start will be used.</li> <li>Missing Stop Month: 'December' will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |

205767

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Laboratory Values

| Hematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hemoglobin | g/dL | | < 8 g/dL | > 13 g/dL |
| Platelet Count | GI/L or x10 <sup>9</sup> / L | | < 80 GI/L | > 500 GI/L |
| WBC Count | GI/L or x10 <sup>9</sup> / L | | < LLRR | > 5x ULRR |
| Neutrophils | GI/L or x10 <sup>9</sup> / L | | < 0.5 GI/L | |
| Lymphocytes | GI/L or x10 <sup>9</sup> / L | | < 0.5x LLRR | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | < 30 g/L | > 55 g/L |
| AST (SGOT) | U/L | | | >= 3x ULRR |
| ALT (SGPT) | U/L | | | >= 3x ULRR |
| Total billirubin | Umol/L | | | >= 2x ULRR |
| Potassium | mmol/L | | > 0.5 mmol/L below LLRR | > 1.0 mmol/L above<br>ULRR |
| Sodium (serum) | mmol/L | | < 130 mmol/L | > 150 mmol/L |

| Iron Parameters | | | | |
|---|---|---|---|---|
| Toot Analyte | Units | Cotomomi | Clinical Concern Range | |
| Test Analyte | Units | Category | Low Flag (< x) | High Flag (>x) |
| Serum ferritin | ug/l | | < 100 ug/l | > 800 ug/l |
| TSAT | Percent | | <15% | > 40% |

# 10.8.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <= 80 mmHg | >= 160 mmHg |
| Diastolic Blood Pressure | mmHg | <= 50 mmHg | >= 100 mmHg |
| Heart Rate | bpm | <= 40 bpm | >= 110 bpm |

Note:

At visits where BP and HR are assessed in triplicate, the average of the 3 values will be used to assess PCI criteria.

205767

10.8.3. FBF

| Agent | Units | Clinical Concern Range | | | |
|--------|----------|------------------------|-------|-----------|------------|
| | | FBF Infused Arm | | FBF Non-I | nfused Arm |
| | | Lower | Upper | Lower | Upper |
| Saline | mL/min | 0.01 | 15.0 | 0.01 | 15.0 |
| ACH | μg/min | 0.01 | 150.0 | 0.01 | 30.0 |
| SNP | μg/min | 0.01 | 150.0 | 0.01 | 30.0 |
| LNMMA | µmol/min | 0.01 | 15.0 | 0.01 | 15.0 |

# 10.8.4. PWV

| PWV Parameter | Units | Clinical Cor | ncern Range |
|----------------------------------------|-------|--------------|-------------|
| | | Lower | Upper |
| Average Systolic BP (Seated & Supine) | mmHg | <= 80 mmHg | >= 160 mmHg |
| Average Diastolic BP (Seated & Supine) | mmHg | <= 50 mmHg | >= 100 mmHg |
| Central Systolic Pressure | mmHg | <= 80 mmHg | >= 160 mmHg |
| Central Diastolic Pressure | mmHg | <= 50 mmHg | >= 100 mmHg |
| Mean Arterial Pressure | mmHg | <= 40 mmHg | >= 200 mmHg |
| Central Pulse Pressure | mmHg | <= 10 mmHg | >= 200 mmHg |
| Peripheral Pulse Pressure | mmHg | <= 10 mmHg | >= 200 mmHg |
| Central Augmentation Pressure | mmHg | <= -50 mmHg | >= 100 mmHg |
| Central Augmentation Index | % | -30 | 60 |
| Heart Rate | bpm | <= 40 bpm | >= 110 bpm |
| Aortic Tr | msec | <=0 msec | >=1000 msec |
| Carotid to Femoral Distance | mm | <= 200 mm | >= 1500 mm |
| Pulse Wave Velocity | msec | <= 2 msec | >= 35 msec |
| Notch to Carotid Distance | mm | <= 10 mm | >= 200 mm |
| Notch to Femoral Distance | mm | <= 200 mm | >= 1500 mm |

# 10.9. Appendix 9: Abbreviations & Trademarks

# 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACH | Acetylcholine, |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIX | Augmentation Index |
| BP | Blood Pressure |
| CDISC | Clinical Data Interchange Standards Consortium |
| CKD | Chronic Kidney Disease |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FBF | Forearm Blood Flow |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FPD | Future Pipeline Discovery |
| GSK | GlaxoSmithKline |
| HR | Heart Rate |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| L-NMMA | L-N <sup>G</sup> -monomethyl arginine citrate |
| PCI | Potential Clinical Importance |
| PCPS | Projects, Clinical Platforms, and Sciences |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PDPP | Pharmacodynamic Per Protocol |
| PP | Per Protocol |
| PWV | Pulse Wave Velocity |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| rhEPO | Recombinant Human Erythropoietin |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SNP | Sodium Nitroprusside |
| SOP | Standard Operation Procedure |
| SRM | Study Reference Manual |
| TFL | Tables, Figures & Listings |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

# 10.10. Appendix 10: List of Data Displays

## 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables |
|------------------|-------------|
| Study Population | 1.1 to 1.6 |
| Safety | 2.1 to 2.9 |
| Pharmacodynamic | 3.1 to 3.10 |
| Section | Listings |
| ICH Listings | 1 to 16 |
| Other Listings | 17 to 20 |

# 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Table | Listing |
|-----------------|----------------|----------------|
| Safety | SAFE1 | - |
| Pharmacodynamic | PD_T1 to PD_T5 | PD_L1 to PD_L2 |

## NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 10.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

205767

# 10.10.4. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject Disposition | | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Status and Subject Disposition for the Study Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| 1.3. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.4. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.5. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.6. | Safety | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

# 10.10.5. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laboratory: Chemistry | | | | | |
| 2.1. | Safety | SAFE1 | Summary of Chemistry lab values | ICH E3 | SAC |
| 2.2. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC |
| Laboratory: Hematology | | | | | |
| 2.3. | Safety | SAFE1 | Summary of Hematology Values | ICH E3 | SAC |
| 2.4. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
205767

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laboratory: Other Screening Tests | | | | | |
| 2.5. | Safety | SAFE1 | Summary of other screen test lab values | ICH E3 | SAC |
| ECG | ECG | | | | |
| 2.6. | Safety | SAFE1 | Summary of ECG Values | IDSL | SAC |
| 2.7. | Safety | EG2 | Summary of Change from Baseline in ECG Values | IDSL | SAC |
| Vital Si | Vital Signs | | | | |
| 2.8. | Safety | SAFE1 | Summary of Vital Signs | ICH E3 | SAC |
| 2.9. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |

## 10.10.6. Pharmacodynamic Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Primary Endpoint | | | | |
| 3.1. | PDPP | PD_T1 | Summary of Forearm Blood Flow Ratio in Response to Acetylcholine | | SAC |
| 3.2. | PDPP | PD_T2 | Summary of Change in Forearm Blood Flow Ratio (Day 1 to Day 42), Acetylcholine | | SAC |
| Princip | Principle Secondary Endpoint | | | | |
| 3.3. | PDPP | PD_T3 | Summary of Change in Absolute Forearm Blood Flow (Day 1 to Day 42), Acetylcholine | | SAC |

205767

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | Secondary Endpoints | | | | |
| 3.4. | PDPP | PD_T2 | Summmary of Change in Forearm Blood Flow Ratio (Day 1 to Day 42), Sodium Nitroprusside | | SAC |
| 3.5. | PDPP | PD_T3 | Summary of Change in Absolute Forearm Blood Flow (Day 1 to Day 42), Sodium Nitroprusside | | SAC |
| 3.6. | PDPP | PD_T2 | Summary of Change in Forearm Blood Flow Ratio (Day 1 to Day 42), L-NMMA | | SAC |
| 3.7. | PDPP | PD_T3 | Summary of Change in Absolute Forearm Blood Flow (Day 1 to Day 42), L-NMMA | | SAC |
| 3.8. | PDPP | PD_T4 | Summary of Augmentation Index and Pulse Wave Velocity | | SAC |
| 3.9. | PDPP | PD_T5 | Summary of Change in Augmentation Index (Day 1 to Day 42) | | SAC |
| 3.10. | PDPP | PD_T5 | Summary of Change in Pulse Wave Velocity (Day 1 to Day 42) | | SAC |

## 10.10.7. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Programming Notes | Deliverable<br>[Priority] | |
| Subject | Subject Disposition | | | | |
| 1. | 1. Screened ES7 Listi | | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | 2. Enrolled ES2 Listing of Reasons for | | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |

| ICH: Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoc | ol Deviations | | | | |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 5. | Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Demog | graphic Charac | teristics | | | |
| 6. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| Prior a | nd Concomitar | nt Medications | | | |
| 7. | Safety | CM10 | Listing of Concomitant Medications | IDSL | SAC |
| 8. | Safety | MH2 | Listing of Medical Conditions | IDSL | SAC |
| Expos | ure | | | | |
| 9. | Safety | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | se Events | | | | |
| 10. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| Seriou | s Adverse Eve | nts | | | |
| 11. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 12. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| All Lab | oratory | | | | |
| 13. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | SAC |
| 14. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |

205767

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | ECG | | | | |
| 15. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| Vital Si | gns | | | | |
| 16. | Safety | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |

## 10.10.8. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Primary Endpoint | | | | |
| 17. | PDPP | PD_L1 | Listing of Forearm Blood Flow | | SAC |
| 18. | PDPP | PD_L2 | Listing of All Forearm Blood Flow Data for Participants with Any Value of Potential Clinical Importance | | SAC |
| Second | lary Endpoint | | | | |
| 19. | PDPP | PD_L3 | Listing of Pulse Wave Velocity and Augmentation Index | | SAC |
| 20. | PDPP | PD_L4 | Listing of All Pulse Wave Velocity and Augmentation Index<br>Data for Participants with Any Value of Potential Clinical<br>Importance | | SAC |

205767

# 10.11. Appendix 11: Example Mock Shells for Data Displays

205767


Example: SAFE1
Protocol: 205767
Population: Safety

Table 2.1
Summary of Lab Values

| | | | Visit | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Treatment | N | | n | Mean | SD | Min | P25 | Median | P75 | Max |
| HGB<br>(g/dL) | Dapro | XXXX | Screening [1] | Xxxx | XX.X | xx.xx | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 1 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Repeat Day 1 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 14 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 28 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 42 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Repeat Day 42 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Follow-up | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | XX |
| | rhEPO | XXXX | Screening [1] | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 1 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Repeat Day 1 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 14 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 28 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Day 42 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Repeat Day 42 | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |
| | | | Follow-up | Xxxx | XX.X | XX.XX | Xx | XX.X | XX.X | XX.X | Xx |

<sup>[1]</sup> Screening is an average of all screening values.

205767

Example: PD T1 Page 1 of n

Protocol: 205767 Population: PDPP

Table 3.1 Summary of Forearm Blood Flow Ratio in Response to Acetylcholine

| Treatment: Daprodustat | | | FBF Con | FBF Control Arm FBF Infuse | | sed Arm | Ratio [1] |
|---|---|---|---|---|---|---|---|
| | Challenge Agent | | Day 1 | Day 42 | Day 1 | Day 42 | |
| | Saline | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 0.834<br>1.65<br>1.0 | 0.834 |
| | 7.5 ug | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 0.834<br>1.65<br>1.0 | |
| | 15 ug | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 1.75<br>0.834<br>1.65 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 0.834<br>1.65<br>1.0 | 0.834 |

<sup>[1]</sup> The Day 42 ratio is calculated by taking the subject's Day 42 treatment (infused) arm and dividing by the Day 42 non-treatment (control) arm value. The Day 1 ratio is calculated by taking the subject's Day 1 treatment (infused) arm and dividing by the Day 1 non-treatment (control) arm value. The overall ratio is determined by taking the subject's Day 42 ratio and dividing by the Day 1 ratio.

205767

Example: PD\_T2 Page 1 of n

Protocol: 205767 Population: PDPP

Table 3.2 Summary of Change in Forearm Blood Flow (FBF) Ratio (Day 1 to Day 42), Acetylcholine

| Challenge Age | nt | Daprodustat<br>FBF Ratio [1] | | Change in FBF Ratio [2] |
|---|---|---|---|---|
| Saline | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 |
| 7.5 ug | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 |
| 15 ug | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 | 3<br>1.75<br>0.834<br>1.65<br>1.0 |

<sup>[1]</sup> The Day 42 ratio is calculated by taking the subject's Day 42 treatment (infused) arm and dividing by the Day 42 non-treatment (control) arm value. The Day 1 ratio is calculated by taking the subject's Day 1 treatment (infused) arm and dividing by the Day 1 non-treatment (control) arm value. The overall ratio is determined by taking the subject's Day 42 ratio and dividing by the Day 1 ratio.

[2] The FBF ratio difference between Daprodustat and rhEPO.

Example: PD T3

Example: PD\_T3
Protocol: 205767
Population: PDPP

Table 3.3 Summary of Change in Absolute FBF (Day 1 to Day 42), Acetylcholine

205767


| Treatment | Challenge Agent | N V | sit | n | Mean | SD | Median | Min. | Max. | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dapro | Saline | | G. Day<br>G. Day | | | | 1.06 | | | 0.7 | 1.7<br>0.5 |
| | 7.5 ug | | G. Day<br>G. Day | | | | 1.06<br>-0.17 | | | 0.7<br>-0.6 | 1.7<br>0.5 |
| | 15 ug | | G. Day<br>G. Day | | | | 1.06<br>-0.17 | 6.69<br>5.72 | | 0.7<br>-0.6 | 1.7<br>0.5 |
| | 30 ug | | G. Day<br>G. Day | | | | 1.06<br>-0.17 | | | 0.7<br>-0.6 | 1.7<br>0.5 |
| rhEPO | Saline | | G. Day<br>G. Day | | | | 1.06<br>-0.17 | 6.69<br>5.72 | | 0.7<br>-0.6 | 1.7<br>0.5 |
| | 7.5 ug | | G. Day<br>G. Day | | | | 1.06<br>-0.17 | 6.69<br>5.72 | | 0.7<br>-0.6 | 1.7<br>0.5 |
| | 15 ug | | G. Day<br>NG. Da | | 2 | | 1.06<br>-0.17 | 6.69<br>5.72 | | 0.7<br>-0.6 | 1.7<br>0.5 |
| | 30 ug | | G. Day | | | | 1.06<br>-0.17 | 6.69<br>5.72 | | 0.7<br>-0.6 | 1.7<br>0.5 |

Example: PD\_T4
Protocol: 205767


Population: PDPP

Table 3.8 Summary of Augmentation Index and Pulse Wave Velocity

| Treatment | | | Day 1 | Day 42 |
|---|---|---|---|---|
| Dapro | Augmentation<br>Index | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 3<br>25.0<br>0.15<br>25.5<br>20<br>30 | 0.15<br>25.5 |
| | Pulse Wave<br>Velocity | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 3<br>7.75<br>0.834<br>6.65<br>7.0<br>9.5 | 0.834<br>6.65<br>7.0 |
| rhEPO | Augmentation<br>Index | n<br>Mean<br>SD<br>Median<br>Min.<br>Max | 1<br>25.0<br>0.15<br>25.5<br>20<br>30 | |

Example: PD\_T5
Protocol: 205767


Population: PDPP

Table 3.9
Summary of Change in Augmentation Index and Pulse Wave Velocity (Day 1 to Day 42)

| Treatment | | N | Visit | n M | lean ( | SD M | Median M | in. Ma | х. |
|---|---|---|---|---|---|---|---|---|---|
| Dapro | Augmentation Index | 4 | AVG. Day 1<br>AVG. Day 42 | 3<br>3 | 24.0<br>-2.0 | 6.69<br>5.72 | 24.5 | 20<br>-2 | 30<br>-3 |
| | Pulse Wave Velocity | 4 | AVG. Day 1<br>AVG. Day 42 | 3 | 7.75<br>-0.50 | 6.695<br>5.722 | 7.50<br>1.50 | 6.0<br>-0.5 | 9.5<br>0.5 |
| rhEPO | Augmentation Index | 4 | AVG. Day 1<br>AVG. Day 42 | 3 | | 6.69<br>5.72 | 24.5<br>-2.5 | 20<br>-2 | 30<br>-3 |
| | Pulse Wave Velocity | 4 | AVG. Day 1<br>AVG. Day 42 | 3 | 7.75<br>-0.50 | 6.695<br>5.722 | 7.50<br>1.50 | 6.0<br>-0.5 | 9.5<br>0.5 |

Example : PD\_L1
Protocol : 205767
Population : PDPP


205767

Listing 17
Listing of Forearm Blood Flow

| Treatment | Unique Subject<br>Id./<br>Subject Id. | Age<br>(YEARS)/<br>Sex/<br>Race<br>Detail | Visit | Challeng<br>e Agent | Challenge<br>Agent<br>Dose | Infusion<br>Drug Unit | Avg.Infus<br>ed Arm | Avg.Non-<br>infused<br>Arm | FBF<br>Rati<br>o |
|---|---|---|---|---|---|---|---|---|---|
| Dapro | PPD | 65/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | Day1 | 1 | 1 | mL/min | 1.2 | 1.3 | 1.22 |
| | | | POST<br>DOSE | 2 | 7.5 | μg/min | 1.4 | 1.01 | 1.33 |
| rhEPO | PPD | 65/<br>F/<br>MIXED<br>RACE | PRE-<br>DOSE | 1 | 1 | mL/min | 1.2 | 1.3 | 1.22 |

Example : PD\_L2
Protocol : 205767
Population : PDPP


Listing of All Forearm Blood Flow Data for Participants with Any Value of Potential Clinical Importance

| Treatment | Arm | Unique Subject<br>Id./<br>Subject Id. | Age<br>(YEARS)/<br>Sex/<br>Race<br>Detail | Visit/<br>Date[Time] | Saline<br>(mL/min) | Ach<br>( <b>µg/min)</b> | SNP<br>( <b>µg/min)</b> | LNMMA<br>(µmol/min) |
|---|---|---|---|---|---|---|---|---|
| Dapro | FBF - infused arm | PPD | 65/<br>F/<br>ASIAN - | PRE-DOSE/<br>2002-01-01<br>T14:00 | хх Н | xx L | хх Н | хх Н |
| | | | JAPANESE<br>HERITAGE | POST DOSE/<br>2002-01-01<br>T14:00 | xx H | xx L | хх Н | хх Н |
| | FBF - non infused arm | PPD | 65/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | PRE-DOSE/<br>2002-01-01<br>T14:00 | хх Н | xx L | хх Н | xx<br>H |
| rhEPO | FBF - infused arm | PPD | 65/<br>F/<br>MIXED<br>RACE | PRE-DOSE/<br>2002-01-01<br>T14:00 | хх Н | xx L | хх Н | хх Н |
| Note: (PCI) | Potential Clinio | cal Importance 1 | Flag: L=Lov | w, H=High | | | | |
| Example | : PD L3 | | | | | | Page 1 | of n |

205767

Protocol : 205767
Population : PDPP

Listing 19

## Listing of Pulse Wave Velocity and Augmentation Index

| Treatment | Unique Subject<br>Id./<br>Subject Id. | Age<br>(YEARS)/<br>Sex/<br>Race Detail | Visit/Planned<br>Time/<br>ECG Date[Time] | Pulse wave<br>velocity test<br>(unit) | Pulse<br>wave<br>result |
|---|---|---|---|---|---|
| Dapro | PPD | 65/<br>F/<br>ASIAN - JAPANESE<br>HERITAGE | Day1/PRE-<br>DOSE/<br>2002-01-01<br>T14:00 | Central<br>Diastolic BP<br>(mmHg) | xx |
| | | | POST DOSE/<br>2002-01-01<br>T14:00 | Central<br>Diastolic BP<br>(mmHg) | xx |
| rhEPO | PPD | 65/<br>F/<br>MIXED RACE | PRE-DOSE/<br>2002-01-01<br>T14:00 | Central<br>Diastolic BP<br>(mmHg) | xx |

Example : PD\_L4


205767

Protocol : 205767
Population : PDPP

Listing 20

Listing of All Pulse Wave Velocity and Augmentation Index Data for Participants with Any Value of Potential Clinical Importance

| Treatment | Unique Subject<br>Id./<br>Subject Id. | Age<br>(YEARS)/<br>Sex/<br>Race<br>Detail | Visit/Plan<br>ned<br>relative<br>Time/<br>Date[Time] | Central<br>Diastoli<br>c BP<br>(mmHg) | Central<br>Systoli<br>c BP<br>(mmHg) | Heart<br>Rate<br>(bpm) | Pulse<br>Wave<br>Velocit<br>Y |
|---|---|---|---|---|---|---|---|
| Dapro | PPD | 65/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | Day1/PRE-<br>DOSE/<br>2002-01-01<br>T14:00 | xx H > | xx L | хх Н | хх Н |
| rhEDO | | | POST DOSE/<br>2002-01-01<br>T14:00 | xx H > | xx L | хх Н | хх Н |
| rhEPO | PPD | 65/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | PRE-DOSE/<br>2002-01-01<br>T14:00 | xx H > | xx L | хх Н | XX<br>H |

Note: (PCI) Potential Clinical Importance Flag: L=Low, H=High

## Signature Page for 205767 TMF- 2204610 v 1.0

| Reason for signing: Approved | Name: PPD Role: Author |
|---|---|
| | Date of signature: 10-Nov-2020 13:46:45 GMT+0000 |
| Reason for signing: Approved | Name: PPD |
| | Role: Approver |
| | Date of signature: 10-Nov-2020 13:59:49 GMT+0000 |

Signature Page for TMF-2204610 v1.0